CLINICAL TRIAL: NCT07041333
Title: The Effect Of Methylphenıdate Treatment On Neuroınflammatıon Levels In Chıldren Wıth Attentıon Defıcıt Hyperactıvıty Dısorder
Status: Completed | Type: Observational
Sponsor: Enes Faruk ALTUNKILIÇ (Other)
Responsible Party: Sponsor-Investigator, Enes Faruk ALTUNKILIÇ, Child and adolescent psychiatrist, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Other Study IDs: 2025-04-11; Ethics Committee (Other: akırköy Ptof. Dr. Sadi Konuk Training and Research Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: methylphenidate; Attention Deficit Hyperactivity Disorder; ADHD; neuroinflammation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patient group with attention deficit and hyperactivity disorder. The group planned to start methylphenidate treatment independent of the study

SUMMARY:
The aim of this study was to investigate the effect of treatment of ADHD with methylphenidate on neuroinflammation by examining the levels of Interleukin-6 (IL-6), S100B, Claudin-5 in serum samples of patients who were diagnosed with attention deficit hyperactivity disorder (ADHD) and started or planned to start methylphenidate for treatment as per routine, at month 0 before the initiation of methylphenidate treatment and at month 3 after the initiation of treatment.

DETAILED DESCRIPTION:
After informed consent, a structured clinical interview for DSM-5-TR will be conducted using the "Emotional Disorders and Schizophrenia Form for School-Age Children - Current and Lifetime Form DSM-5 - Turkish Adaptation (ÇDŞG-ŞY-DSM-5-T)". The "Sociodemographic and Clinical Data Form" created by the researchers will be completed to obtain sociodemographic and clinical data for the participants. The "Conners Parent Rating Scale-Revised Short Form" and "Conners Teacher Rating Scale-Revised Short Form" will be administered to the group diagnosed with ADHD to determine the severity of the disease, symptoms, and predominant subtypes. After the diagnosis is made and evaluated according to the exclusion criteria, peripheral venous blood will be collected in yellow-capped tubes between 9 and 12 a.m. after a 10-12 hour fast, prior to the routine planned methylphenidate treatment. After being left at room temperature for 10-20 minutes, the blood will be centrifuged at 3000 RPM for 20 minutes, and the serum portion will be collected into Eppendorf tubes and stored at -80 degrees until the samples are analyzed. Three months after starting treatment, blood will be collected and stored in the same manner. After all samples have been collected, the serum samples will be analyzed in a single batch for Interleukin-6 (IL-6), S100B, and Claudin-5 levels using human ELISA kit protocols at the Medical Biochemistry Laboratory of Bakırköy Dr. Sadi Konuk Training and Research Hospital by biochemistry specialist Dr. Hacer Eroğlu İçli. Three months after the start of treatment, the Conners Parent Rating Scale - Revised Short Form and the Conners Teacher Rating Scale - Revised Short Form will be administered again.

ELIGIBILITY:
Inclusion Criteria:

1. According to DSM-5 TR, the participant must have a diagnosis of "Attention Deficit Hyperactivity Disorder" and have started/be planning to start routine methylphenidate treatment.
2. The participant must be between 6 and 11 years of age.
3. The participant must agree to participate in the study after being informed about it.

Exclusion Criteria:

1. The presence of a psychiatric disorder diagnosis other than Attention Deficit Hyperactivity Disorder
2. Having a diagnosis of Attention Deficit Hyperactivity Disorder but not planning to start methylphenidate
3. Being under 6 years of age or over 11 years of age
4. Having organic brain damage, mental retardation, autism spectrum disorder, neurological disease, or a physical illness that affects neurocognitive functions
5. History of alcohol and/or psychoactive substance use
6. Presence of ongoing active infection, allergic disease, and chronic illness
7. Previous use of psychiatric medication.
8. Presence of chronic illness
9. Regular use of medication

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who applied to Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, diagnosed with Attention Deficit Hyperactivity Disorder, deemed suitable for methylphenidate treatment, and for whom methylphenidate treatment is planned, have been referred to us.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-10-19 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospita, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The participants' age, scores of the clinical scales examined in the study, and levels of serum samples will be shared. In other words, the necessary data relevant to the purpose of the study will be shared.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Hogasen AK, Hestdal K, Abrahamsen TG. Granulocyte-macrophage colony-stimulating factor, but not macrophage colony-stimulating factor, suppresses basal and lipopolysaccharide-stimulated complement factor production in human monocytes. J Immunol. 1993 Sep 15;151(6):3215-24. PMID 7690797
- [Background] Leung AK, Hon KL. Attention-Deficit/Hyperactivity Disorder. Adv Pediatr. 2016 Aug;63(1):255-80. doi: 10.1016/j.yapd.2016.04.017. No abstract available. PMID 27426904
- [Background] Kul M, Unal F, Kandemir H, Sarkarati B, Kilinc K, Kandemir SB. Evaluation of Oxidative Metabolism in Child and Adolescent Patients with Attention Deficit Hyperactivity Disorder. Psychiatry Investig. 2015 Jul;12(3):361-6. doi: 10.4306/pi.2015.12.3.361. Epub 2015 Jul 6. PMID 26207130
- [Background] Koc S, Guler EM, Derin S, Gultekin F, Aktas S. Oxidative and Inflammatory Parameters in Children and Adolescents With ADHD. J Atten Disord. 2023 Jun;27(8):880-886. doi: 10.1177/10870547231159907. Epub 2023 Mar 6. PMID 36879528

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially, 42 patients were enrolled in the study. During the follow-up period, a new patient was recruited to replace each patient who withdrew before completing the study. Consequently, a total of 57 patients were enrolled, and 15 patients withdrew from the study for various reasons.
Period: Overall Study
Arm/Group | Patient Group
Started | 57
Completed | 42
Not Completed | 15
Not completed — Lost to Follow-up | 7
Not completed — Side effect | 3
Not completed — Medication refusal by the child. | 3
Not completed — Medication refusal by the family. | 1
Not completed — The family's request to obtain a second medical opinion. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patient Group
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.32 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 42
kilogram (kg) [Mean (Standard Deviation); unit: kilogram (kg)] | 27.6 (7.22)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — BMI-for-age Z-score (age- and sex-standardized). Z=0 is the reference mean; +1 and +2 indicate 1 and 2 SD above the mean, respectively; negative values indicate below-average BMI. Higher Z-scores indicate higher BMI. Clinically relevant cut points: Z ≥ +2 obesity; Z ≥ +1 overweight; Z ≤ -2 underweight/thinness; Z ≤ -3 severe thinness.
  kg/m² | 16.5 (1.93)
Body Mass Index (BMI) z-score [Mean (Standard Deviation); unit: z-score] | 0.13 (0.84)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 128 (0.11)
School year (year(s)) [Median (Inter-Quartile Range); unit: years] | 2.5 [1.25 to 4]
ADHD presentation type [Count of Participants; unit: Participants]
  Combined presentation | 29
  Predominantly inattentive presentation | 9
  Predominantly hyperactive-impulsive presentation | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in IL-6 Marker Level
Description: Interleukin-6 (IL-6) level was measured according to the human ELISA kit protocol. Serum samples from 42 patients were compared immediately before and after 3 months of treatment. IL-6 was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E0090Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-IL-6 antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Patient Group
Number analyzed (Participants) | 42
ng/L
  IL-6 (before starting treatment) | 113.89 (121.27)
  IL-6 (after starting treatment) | 103.45 (101.62)
Statistical Analysis 1: Comparison: Patient Group; Test type: Superiority; p = 0.014, t-test, 2 sided; Paired-samples t-test

2. Primary Outcome: Change in S100B Marker Level
Description: S100 Calcium Binding Protein B (S100B) level was measured according to the human ELISA kit protocol. Serum samples from 42 patients were compared immediately before and after 3 months of treatment. S100B was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E3887Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-S100B antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Patient Group
Number analyzed (Participants) | 42
ng/L
  S100B (before starting treatment) | 871.13 [582.27 to 1185.95]
  S100B (after starting treatment) | 758.13 [507.67 to 1031.77]
Statistical Analysis 1: Comparison: Patient Group; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in the Level of Claudin-5 Marker
Description: Claudin 5 level was measured according to the human ELISA kit protocol. Serum samples from 42 patients were compared immediately before and after 3 months of treatment. Claudin 5 was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E2303Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-Claudin 5 antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Patient Group
Number analyzed (Participants) | 42
ng/L
  Claudin 5 (before starting treatment) | 206.52 [118.29 to 473.93]
  Claudin 5 (after starting treatment) | 181.76 [124.32 to 367.88]
Statistical Analysis 1: Comparison: Patient Group; Test type: Superiority; p = 0.175, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients diagnosed with attention deficit hyperactivity and planned to receive methylphenidate treatment were included in the study. Patients eligible for methylphenidate treatment due to indication were included. Therefore, there were no patients at risk of death or serious adverse events.
Arm/Group | Patient Group
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 30/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Group (N=57)
loss of appetite (General disorders) | 22 — This adverse effect was observed transiently within the first 3 months in 7 children, whereas it persisted throughout the 3-month period in the other 15 children.
Weight loss (General disorders) | 1 — This adverse effect was observed throughout the 3-month period in one child.
Headache (General disorders) | 3 — This adverse effect was observed transiently within the first 3 months in three children.
Dizziness (General disorders) | 1 — This adverse effect was observed transiently within the first 3 months in one child.
abdominal pain (General disorders) | 4 — This adverse effect was observed transiently within the first 3 months in four children.
Nausea (General disorders) | 4 — This adverse effect was observed transiently within the first 3 months in four children.
Agitation (General disorders) | 1 — This adverse effect was observed transiently within the first 3 months in one child.
Extreme stagnation (General disorders) | 7 — This adverse effect was observed transiently within the first 3 months in seven children.
Chest pain (General disorders) | 1 — This adverse effect was observed transiently within the first 3 months in one child.
Tachycardia (General disorders) | 1 — This adverse effect was observed transiently within the first 3 months in one child.
Difficulty falling asleep at night (General disorders) | 4 — This adverse effect was observed transiently within the first 3 months in three children, whereas it persisted throughout the 3-month period in one child.
Blurred vision (General disorders) | 1 — This adverse effect was observed transiently within the first 3 months in one child.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT07041333/Prot_SAP_ICF_001.pdf